CLINICAL TRIAL: NCT02109627
Title: Phase Ib Study of Ficlatuzumab With High Dose Cytarabine (HiDAC) in Relapsed and Refractory AML
Brief Title: Ficlatuzumab With High Dose Cytarabine in Relapsed and Refractory AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: C. Babis Andreadis (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, C. Babis Andreadis, Associate Professor of Clinical Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 139510; NCI-2015-00749 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-01-23; First posted 2014-04-10 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Ficlatuzumab; High Dose Cytarabine; antibody
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ficlatuzumab; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ficlatuzumab, Cytarabine (Experimental): Ficlatuzumab 5-20 mg/kg; intravenous; Days 0, 14, 28, 42; Number of cycles: until progression or unacceptable toxicity develops.
  Cytarabine 2 g/m2; intravenous; Days 2-7; Number of cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: Ficlatuzumab; Drug: Cytarabine

INTERVENTIONS:
Drug: Ficlatuzumab — 5-20 mg/kg; intravenous; Days 0, 14, 28, and 42. Number of cycles: until progression or unacceptable toxicity develops.
Drug: Cytarabine — 2 g/m2; intravenous; Days 2-7; Number of cycles: until progression or unacceptable toxicity develops.
  Other Names: HiDAC

SUMMARY:
The purpose of this study is to see if ficlatuzumab when combined with cytarabine, a standard treatment for AML, is safe to give to patients and to determine the best dose to give. The study doctors want to see what effects, good and/or bad, the study drug has on subjects and their AML. The study will look at what side effects subjects may have and how subjects feel after receiving the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory AML as defined by one of the following criteria:

  1. First relapse within 12 months after date of first Complete Response (CR) or complete repsonse with incomplete hematologic recovery (CRi)
  2. Persistent AML documented by bone marrow biopsy at least 28 days after day 1 of the first induction cycle of cytotoxic chemotherapy
  3. Hypercellular bone marrow with greater than 20% cellularity and 10% blasts at least 14 days after first induction cycle day 1
* Age >=18
* Prior induction therapy had to include no more than two cycles of cytotoxic chemotherapy and at least one induction cycle must have consisted of an anthracycline or anthracenedione and cytarabine combination with a reasonable schedule/dose according to the discretion of the investigator
* Histologically confirmed AML by hematopathology review performed within four weeks prior to study entry
* Ejection fraction >=40% by transthoracic echocardiogram or radionuclide ventriculogram, i.e. multigated acquisition (MUGA) scan
* Treatment for non-hematologic malignancy greater than 6 months prior to enrollment is acceptable.
* Transplantation for AML (allogeneic or autologous) allowed unless within 90 days of study entry
* No active graft versus host disease (GVHD) or immunosuppression for prevention or treatment of GVHD within two weeks of study entry
* Prior treatment of myelodysplastic syndrome or myeloproliferative neoplasm with hypomethylating agent acceptable.
* Cytoreduction therapy with plasmapheresis or hydroxyurea acceptable.
* Females must have a negative serum pregnancy test 24 hours prior to the start of treatment or be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months)
* Adequate liver function as defined by total bilirubin ≤ 2.0 mg/dL (≤ 3.0 mg/dL for patients with known Gilbert's syndrome) and aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 3 times upper limit of normal, unless these are thought to be due to AML
* Adequate renal function with creatinine ≤ 2.0 mg/dL
* The effects of ficlatuzumab on the developing human fetus are unknown. For this reason and because cytarabine is pregnancy category D, women of child-bearing potential and men must agree to use adequate contraception: hormone, barrier method of birth control, or abstinence prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and at least one month after completion of study drug administration.
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Acute promyelocytic leukemia (FAB M3 AML)
* More than 2 cycles of prior induction therapy for AML
* Allogeneic or autologous transplant for AML with infusion of stem cells within 90 days of study entry or on active immunosuppressive therapy for graft versus host disease (GVHD) within 2 weeks before study entry
* Cytarabine containing regimen in excess of 2 g/m2/day within 6 months of study entry
* Chemotherapy, radiation, or immunotherapy, within 2 weeks prior to study entry, other than those specified in the inclusion criteria (hydroxyurea and hypomethylating agents)
* Known active HIV, hepatitis B or C or infection. Exception for patients with hepatitis B on antivirals and low viral load, to be determined at the discretion of the investigator.
* Uncontrolled infection
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Active second malignancy that in the opinion of the PI may interfere with or be adversely affected by this treatment.
* Prior exposure to the investigational agent or anti-c-Met, anti-HGF or anti-VEGF directed therapy within six months prior to study entry
* Prior grade 4 toxicity attributed to cytarabine
* Known or suspected drug sensitivity to cytarabine or the investigational agent ficlatuzumab
* Inability to provide consent
* Pregnant women are excluded from this study because the effect of ficlatuzumab on the developing fetus remains unknown and that cytarabine is a pregnancy risk category D drug with known teratogenic or abortifacient effects. Because of the potential adverse events in nursing infants secondary to treatment of the mother with ficlatuzumab and cytarabine, breastfeeding should be discontinued while on study. Patients who become pregnant while on study will be removed from the study once the pregnancy is confirmed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) for ficlatuzumab when administered with HiDAC | Up to 2 years
Maximum Tolerated Dose (MTD) for ficlatuzumab when administered with HiDAC | Up to 2 years

SECONDARY OUTCOMES:
Preliminary activity of ficlatuzumab in combination with HiDAC in patients with relapsed or refractory AML | Up to 2 years
Functional status for patients receiving ficlatuzumab and HiDAC | Up to 2 years
Quality of life for patients receiving ficlatuzumab and HiDAC | Up to 2 years

OTHER OUTCOMES:
Overall survival of patients receiving ficlatuzumab in combination with HiDAC | Up to 2 years
Candidate biomarkers for response to combination therapy | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Andreadis, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No